CLINICAL TRIAL: NCT05795010
Title: Observation of MRD Detection for Preoperative Sensitivity and Postoperative Positive Rate in Common Risk Stage II Colorectal Cancer
Brief Title: MRD Test in Common Risk Stage II Colorectal Cancer
Acronym: HuaMC-1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-174
Record Dates: First submitted 2023-03-07; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Stage II Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Tumor tissue and venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MRD test — ctDNA detection based on tumor whole exon sequencing
  Other Names: ctDNA test

SUMMARY:
Patients with colorectal cancer who were confirmed as stage II general risk type in the postoperative pathological report began to be enrolled. Observe the sensitivity of the detection of micro-MRD before operation and the postoperative positive rate of this type of patients.

DETAILED DESCRIPTION:
This observation part is about the patients with general risk stage II colorectal cancer who have received R0 resection after screening by nanofiltration criteria. Twenty milliliters of venous blood samples were reserved before surgery, and tumor tissue samples were reserved within 30 minutes in vitro during surgery. After the pathological diagnosis of the patients after surgery, they began to be enrolled. To observe the sensitivity of MRD detection in preoperative diagnosis of patients with general risk stage II colorectal cancer, and to study its positive rate one month and three months after operation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75;
* Pathologically confirmed rectal adenocarcinoma;
* Pathological differentiation is highly or moderately differentiated;
* The pathological stage was pT3N0, that is, invasion of the proper muscular layer of the intestinal wall without lymph node metastasis;
* No new adjuvant treatment before operation
* There was no vascular infiltration and nerve infiltration in postoperative pathology;
* No preoperative intestinal obstruction or tumor site perforation;
* No postoperative pathological margin was positive or unknown;
* The distance between the pathological cutting edge and the tumor was more than 1 cm;
* Invasion of mesentery of intestinal wall ≤ 2mm;
* More than 12 lymph nodes were submitted for examination;
* Nonlocal recurrence and distant metastasis;
* No multiple primary carcinoma of colon and rectum;
* Physical condition score PS ≤ 2 points;
* Patients and their families can understand and are willing to participate in this study and provide written informed consent.

Exclusion Criteria:

* Multiple intestinal carcinomatosis
* Previous history of malignant tumor,
* There are concurrent malignant tumors in the whole body except for colorectal cancer
* Colorectal cancer with preoperative anti-tumor treatment
* Pregnant or lactating women
* There are serious complications during or after operation, affecting the prognosis
* Hepatitis B or Hepatitis C antibody positive
* HIV antibody positive
* Other diseases considered by the research doctor to affect the prognosis and survival
* Other conditions that the research doctor believes are not consistent with this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Preoperative venous blood and intraoperative tumor tissue samples were reserved for patients with colorectal cancer who were estimated as stage II general risk type by pelvic magnetic resonance imaging. Patients with colorectal cancer who were confirmed as stage II general risk type in the postoperative pathological report began to be enrolled
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-03-30 (Estimated); Primary Completion 2023-04-10 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Positive rate of preoperative MRD test | six months
  To observe the positive rate of preoperative MRD detection for stage II colorectal cancer

SECONDARY OUTCOMES:
Positive rate of MRD test 1 month and 3 months after operation | nine months
  Observe the positive rate of MRD detection at 1 month and 3 months after operation for stage II colorectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Yongchun Song, MD, Study Chair — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be published anonymously after the end of the study

REFERENCES:
- [Background] Reinert T, Henriksen TV, Christensen E, Sharma S, Salari R, Sethi H, Knudsen M, Nordentoft I, Wu HT, Tin AS, Heilskov Rasmussen M, Vang S, Shchegrova S, Frydendahl Boll Johansen A, Srinivasan R, Assaf Z, Balcioglu M, Olson A, Dashner S, Hafez D, Navarro S, Goel S, Rabinowitz M, Billings P, Sigurjonsson S, Dyrskjot L, Swenerton R, Aleshin A, Laurberg S, Husted Madsen A, Kannerup AS, Stribolt K, Palmelund Krag S, Iversen LH, Gotschalck Sunesen K, Lin CJ, Zimmermann BG, Lindbjerg Andersen C. Analysis of Plasma Cell-Free DNA by Ultradeep Sequencing in Patients With Stages I to III Colorectal Cancer. JAMA Oncol. 2019 Aug 1;5(8):1124-1131. doi: 10.1001/jamaoncol.2019.0528. PMID 31070691
- [Background] Romero D. ctDNA guides omission of adjuvant chemotherapy for stage II CRC. Nat Rev Clin Oncol. 2022 Aug;19(8):493. doi: 10.1038/s41571-022-00657-7. No abstract available. PMID 35750857
- [Result] Tie J, Cohen JD, Lahouel K, Lo SN, Wang Y, Kosmider S, Wong R, Shapiro J, Lee M, Harris S, Khattak A, Burge M, Harris M, Lynam J, Nott L, Day F, Hayes T, McLachlan SA, Lee B, Ptak J, Silliman N, Dobbyn L, Popoli M, Hruban R, Lennon AM, Papadopoulos N, Kinzler KW, Vogelstein B, Tomasetti C, Gibbs P; DYNAMIC Investigators. Circulating Tumor DNA Analysis Guiding Adjuvant Therapy in Stage II Colon Cancer. N Engl J Med. 2022 Jun 16;386(24):2261-2272. doi: 10.1056/NEJMoa2200075. Epub 2022 Jun 4. PMID 35657320

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-25): https://cdn.clinicaltrials.gov/large-docs/10/NCT05795010/Prot_SAP_000.pdf